CLINICAL TRIAL: NCT00221039
Title: UVADEX Sterile Solution in Conjunction With the UVAR XTS Photopheresis System as an Interventional Therapy for the Treatment Of CTCL (Mycosis Fungoides) in Patients With TMN Classification Stage 1A, 1B, 2A
Brief Title: Photopheresis as an Interventional Therapy for the Treatment of CTCL (Cutaneous T-Cell Lymphoma, Mycosis Fungoides) Stage 1A, 1B, 2A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Boston Medical Center (Other); University of Pittsburgh (Other); Case Western Reserve University (Other); Vanderbilt University Medical Center (Other); University of Minnesota (Other); Rush University Medical Center (Other); Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECTCL1
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Cutaneous T Cell Lymphoma; Mycosis Fungoides
Keywords: ECP; Photopheresis; CTCL; Cutaneous T Cell Lymphoma; Mycosis Fungoides
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DRUG+ECP (Experimental): UVVADEX +ECP will be administered to patients with CTCL.Duration of Treatment: The study will consist of 2 treatment periods, a 6-month initial period and a 6-month follow-up period where photopheresis therapy may continue.
  Interventions: Drug: Methoxsalen+ECP

INTERVENTIONS:
Drug: Methoxsalen+ECP — UVAdex+ECP will be administered: Treatment consists of two photopheresis treatments on successive days every 4 weeks for six months
  Other Names: Uvadex

SUMMARY:
The study objective is to demonstrate that the UVADEX® Sterile Solution formulation of methoxsalen used in conjunction with the UVAR XTS Photopheresis System can have a clinical effect on the skin manifestations of CTCL (mycosis fungoides) in early stage disease.

DETAILED DESCRIPTION:
Objectives: The study objective is to demonstrate that the UVADEX® Sterile Solution formulation of methoxsalen used in conjunction with the UVAR XTS Photopheresis System can have a clinical effect on the skin manifestations of CTCL (mycosis fungoides) in early stage disease.

Methodology: Single-arm, open-label treatment using UVAR XTS Photopheresis System. Treatment consists of two photopheresis treatments on successive days every 4 weeks for six months. Those patients completing the first 6-month period may be continued on photopheresis for a 6-month follow-up period. Patients who do not respond to photopheresis therapy after 6 months may have concurrent therapy with low dose bexarotene and interferon added as outlined in the protocol.

Number of Patients (Planned and Analyzed): The study plan is for a minimum of 50 patients

Diagnosis and Main Criteria for Inclusion: Male or female patients with CTCL diagnosis of stage IA, IB or IIA with measurable skin lesions (patches or plaques) and a minor blood abnormality. Patients must be refractory to at least one treatment for early stage CTCL such as PUVA, Electron beam, oral steroids, high potency topical steroid, topical nitrogen mustard, methotrexate, interferon, or bexarotene.

Test Product, Dose and Mode of Administration, Batch or Lot Number: UVADEX liquid methoxsalen 20mcg/mL in conjunction with the UVAR XTS Photopheresis System. UVADEX is injected into the photoactivation bag during photopheresis therapy in accordance with the approved drug package insert and UVAR XTS operator's manual. UVADEX dose is less than 200mcg per treatment.

Duration of Treatment: The study will consist of 2 treatment periods, a 6-month initial period and a 6-month follow-up period where photopheresis therapy may continue.

Criteria for Evaluation:

Efficacy: The primary endpoint will be the overall response based on skin-weighted assessment. Secondary endpoints will also include time to response, duration of response, and a "Quality of Life " assessment. The size and number of lymph nodes and flow cytometry analyses will also be considered. Experienced skin observers will perform skin scores on each patient at enrollment. Skin scores will be recorded as the percentage of the patient's body involved with patch or plaque lesions. A successful response to therapy will be patients who have a greater than 50% improvement in skin involvement (PR) or complete skin improvement (CR) without worsening in nodes, blood or visceral organs. Patients with 25%-50% improvement will be considered as minor response (MR), + or - 25% will be SD, and PD will be defined as 25% worsening from baseline.

Safety: Safety is assessed by the incidence and intensity of adverse events, whether clinical or based on laboratory results.

Statistical Methods: The primary endpoint will be the proportion of patients who have CR and PR of their skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients are to be greater than 40 kg body weight.
* Patients must have adequate veins to provide intravenous access.
* Women who are not pregnant, lactating, or of childbearing potential. Lack of childbearing potential was defined as:

  * Being post-menopausal
  * Being surgically sterile
  * Practicing contraception
* Patients with childbearing potential had to have a negative serum human chorionic gonadotropin (HCG) upon entrance into the study.
* Patients must be willing to adhere to the protocol, and sign an Informed Patient Consent Form prior to entry into the study.
* Patients must not be on any other investigational device/drug treatment.
* Patients with the diagnosis of mycosis fungoides (MF) including a skin biopsy consistent with MF (atypical epidermotrophic or folliculocentric T-cells).
* Appropriate staging as IA, IB or IIA : T1 or T2 (patches or plaques) with measurable lesions.

  * IA patients must show evidence of a minor blood abnormality by morphology or laboratory assessment.
  * For IIA patients - clinically significant nodes (1.5 cm) must have lymph node biopsy showing dermatopathic nodes or no involvement.
* Patients must be willing and able to discontinue concomitant medications for MF.
* Patients currently taking the following drugs must discontinue medication prior to enrollment in the trial:

  * Psoralens and ultraviolet A (PUVA) or ultraviolet B (UVB) therapy - 4 weeks
  * Topical nitrogen mustard or other topical chemotherapy - 4 weeks
  * Bexarotene capsules or other systemic biologic agent - 3 weeks washout
  * High dose topical steroids, topical retinoids or immunotherapy - 2 week washout with 1% topical hydrocortisone
  * Oral steroids above 10 mg - 30 day washout, unless patient has Addison's disease or adrenal insufficiency
* Patients must be refractory to at least one of the standard therapies used to treat Stage IA, IB or IIA CTCL such as oral steroids, high-dose topical steroids, mechlorethamine (HN2), bexarotene, PUVA therapy, electron beam radiation, biological response or oral methotrexate.
* Patients must abstain from therapeutic sunbathing, tanning beds, etc. for the duration of the study.

Exclusion Criteria:

* Patients who have MF (T3 cutaneous tumors or T4 exfoliative erythroderma) Stage IIB - IVB, ie. no pathological node or visceral involvement.
* Patients who are unable to tolerate extracorporeal volume loss (e.g., severe cardiac disease or severe anemia or weight < 40 kg).
* Patients with recent (within three months) deterioration of renal function who have a serum creatinine level greater than 3.0 mg/dL.
* Patients with lipemic plasma > 500 ng/dL or uncontrolled diabetes.
* Patients with a history of liver damage (2.5 x normal ALT, AST) or porphyria.
* Patients with positive tests for HIV antibody, hepatitis C virus (HCV) antibody or hepatitis B surface antigen.
* Patients on oral prednisone therapy or full body or high potency topical steroids.
* Women who are pregnant or nursing a child.
* Patients with severe emotional, behavioral or psychiatric problems that, in the opinion of the investigator, would result in poor compliance with the treatment regimen.
* Patients who exhibit idiosyncratic or hypersensitivity reactions to 8-methoxypsoralen compounds, heparin, or citrate.
* Patients with previous exposure to photopheresis therapy.
* Patients who use tanning beds or are receiving phototherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-04-02 (Actual); Primary Completion 2011-04-05 (Actual); Study Completion 2011-04-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the overall response based on skin-weighted assessment. | 6 months
  The overall skin repsonse will be assessed at 6month and will consist of an experts assessment of the % of skin involvement at baseline and 6 months.

SECONDARY OUTCOMES:
Quality of life assessed by questionnaire | 6 months
  A quality of life questionnaire will be completed by the patient at 6 months of treatment and 6 months after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Duvic, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Rush-Presbyterian Hospital, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University Hospital of Cleveland/Case Western Reserve University, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Talpur R, Demierre MF, Geskin L, Baron E, Pugliese S, Eubank K, Zic JA, Miller DR, Tharp M, Bohjanen K, Duvic M. Multicenter photopheresis intervention trial in early-stage mycosis fungoides. Clin Lymphoma Myeloma Leuk. 2011 Apr;11(2):219-27. doi: 10.1016/j.clml.2011.03.003. Epub 2011 Apr 8. PMID 21575927